CLINICAL TRIAL: NCT01863459
Title: Lisdexamfetamine Dimesylate in the Treatment of Adult ADHD With Anxiety Disorder Comorbidity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Anxiety, Attention Deficit and Trauma, Ontario, Canada (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LDX-COMORB-1
Record Dates: First submitted 2013-05-17; First posted 2013-05-29 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder (ADHD) With Co-occuring Anxiety and Depressive Disorders
Keywords: ADHD; ADD; Anxiety; Anxiety Disorders; Depression; Attention; Attention Deficit
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Depressive Disorder; Anxiety Disorders; Depression | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidexamfetamine Dimesylate (Experimental): Lisdexamfetamine dimesylate (Vyvanse) is a central nervous system (CNS) stimulant, approved for the treatment of ADHD Lisdexamfetamine dimesylate is to be started at a dose of 30 mg/day for one week, increased to 50 mg/day for week 2 and to 70 mg/day for week 3. Doses are increased to the maximally tolerated/efficacious dose. Thirty milligrams of Lisdexamfetamine dimesylate per day, is the minimum dose that must be achieved.
  Duration of treatment in this arm is 8 weeks; tablet is taken once per day
  Interventions: Drug: Lisdexamfetamine Dimesylate
- Placebo (Placebo Comparator): Placebo will be dosed in the same fashion as the active intervention - 3 potential dose levels.
  Placebo is taken once per day for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate
  Other Names: Vyvanse
  Arms: Lidexamfetamine Dimesylate
Drug: placebo
  Arms: Placebo

SUMMARY:
1. To evaluate the safety, and efficacy of Lisdexamfetamine dimesylate in the treatment of outpatients with DSM-IV ADHD with anxiety and depressive disorder comorbidity, as well as to evaluate the effects on quality of life .
2. To evaluate the efficacy of Lisdexamfetamine dimesylate in the treatment of anxiety and depressive disorders which commonly occur with ADHD.
3. To examine the potential relationship between telomere length and Adult ADHD with comorbidity and the potential effect of treatment response.
4. To examine the potential associations with specific genes and Adult ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient men and woman aged 18 to 65 years.
2. Patients with a DSM-IV diagnosis of ADHD according to the MINI-Plus, with an ADHD-RS score ≥ 24 and at least one of the following comorbid psychiatric disorders: SP, PDAG, OCD, GAD, MDD or Dysthymia.
3. Patients who qualify for comorbid DSM-IV major depressive disorder - current episode, will be allowed into the study provided that they have a baseline Montgomery Asberg Depression Rating Scale (MADRS) score of less than or equal to 25.
4. The ability to comprehend and satisfactorily comply with protocol requirements.

6. Written informed consent given prior to entering the baseline period of the study.

7. All women of child bearing potential must have a negative screening visit serum or urine pregnancy test and be using adequate contraception for the duration of the study. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices or properly used barrier contraception. Additionally, the use of condoms is suggested as an adjunct to the methods previously addressed to provide additional protection against accidental pregnancy.

8. Concomitant treatment with selective serotonin reuptake inhibitors (SSRI's), serotonin noradrenaline reuptake inhibitors (SNRI's), benzodiazepines, beta-blockers, atypical anti-psychotics, anti-epileptics is allowed, provided the dose has been stable for 8 weeks prior to study entry. Dose changes of allowed concomitant medication should be avoided during the treatment phases of the study.

-

Exclusion Criteria:

1. Patients who currently fulfill criteria for a lifetime history of bipolar disorder, history of drug abuse, a history of schizophrenia or other psychotic disorders, delirium, dementia and amnesic and other cognitive disorders, or are in a current agitated state.
2. Patients with a concurrent AXIS-II, cluster A personality disorder or borderline or antisocial personality disorder.
3. Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviours within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
4. Patients receiving current psychotherapy, including cognitive behavioural therapy for either ADHD or an anxiety or mood disorder, within 4 weeks prior to the baseline period.
5. Patients who, during the course of the study would be likely to require treatment with a prohibited concomitant therapy (please refer to Concomitant Medication section below).
6. Patients who are known to be allergic to amphetamines or components of Lisdexamfetamine dimesylate, have known hypersensitivity or idiosyncrasy to Lisdexamfetamine dimesylate or sympathomimetic amines.
7. Patients with a current seizure disorder, organic brain disorder or history of seizure disorder (except for febrile seizures in childhood).
8. Patients who have thyroid pathology, treatment of which has not been stabilized for at least 3 months.
9. MAO inhibitors within 3 weeks of the start of the baseline.
10. Current use of bupropion or tri-cyclic antidepressants, with the exception of clomipramine.
11. Current use of clonidine, modafinil or atomoxetine.
12. Previous intolerance or failure to respond to an adequate trial of Lisdexamfetamine dimesylate (defined as a minimum of 30mg per day for at least 4 weeks).
13. Current use of any psycho-stimulant, and greater than 2 failed trials using adequate doses of a methylphenidate-based or amphetamine agent.
14. Pregnant or lactating females or if sexually active and of childbearing potential not using adequate methods of birth control. If a subject becomes pregnant during the study she will be discontinued immediately and followed appropriately (at minimum, until the outcome of the pregnancy is determined).
15. Patients who have a history or evidence of a medical condition that would expose them to an increase or significant adverse event or interfere with assessments of safety and efficacy during the course of the trial including: advanced arteriosclerosis, symptomatic cardiovascular disease, moderate to severe hypertension, or other pre-existing cardiac abnormalities or other serious cardiac problems.
16. Patients with a history of Glaucoma.
17. Sleep medications during the study period are excluded with the exception of zopiclone and over-the-counter sleep aids.
18. Patients using any herbal psychoactive treatments, eg; St.John's Wort, Valerian, Kava Kava, or Chamomile Extract within 14 days prior to randomization.
19. Patients who have received electroconvulsive therapy within the previous 6 months.
20. Patients with any condition or on any therapy that in the investigator's opinion or as indicated in the Lisdexamfetamine dimesylate product label, that may pose a risk to the subject or interfere with the study objective.
21. Patients having clinically significant abnormal laboratory or ECG findings not resolved by the baseline examination.

The exclusion criteria must continue to be satisfied in order for the patient to enter the randomization phase at the end of the baseline.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale | Change from Baseline to Week 18
Clinical Global Impression - Improvement Scale (CGI-I) | Change from Week 1 to Week 18

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Change from Baseline to Week 18
the Overall Anxiety Severity and Impairment Scale (OASIS) | Change from Baseline to Week 18
The Weiss Functional Impairment Rating Scale-Self Report (WFIRS-S) | Change from Baseline to Week 18
Barkley Adult ADHD Rating Scale--IV(BAARS-IV) | Change from Baseline to Week 18
Revised Padua Inventory | Change from Baseline to Week 18
The Panic and Agoraphobia Scale (PAS) | Change from Baseline to Week 18
Quick Inventory of Depressive Symptoms (QID-SR-16) | Change from Baseline to Week 18
The Sheehan Disability Scale (SDS) | Change from Baseline to Week 18
GAD-7 | Change from Baseline to Week 18
Social Phobia Inventory (SPIN) | Change from Baseline to Week 18
The Life Events Questionnaire (LEQ) | Visit 2 (Week: Baseline)
The Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline to Week 18
Clinical Global Impression - Severity (CGI-S) | Change from Baseline to Week 18

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Collins, MBChB, FRCPC, Principal Investigator — McMaster University
Locations (1):
- Centre for Anxiety, Attention Deficit and Trauma, Hamilton, Ontario, Canada

REFERENCES:
- See also: Related Info — http://www.anxietyaddtreatment.com